CLINICAL TRIAL: NCT05775822
Title: Coronary Artery Calcium and Cardiovascular Risk Factors Analysis After RT for Breast Cancer. A Gender-based Preventive Medicine Approach
Brief Title: Coronary Artery Calcium and Cardiovascular Risk Factors Analysis After RT or Breast Cancer
Acronym: RadioTherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Istituto Europeo di Oncologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CCM 1505
Record Dates: First submitted 2023-02-17; First posted 2023-03-20 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Coronary Artery Disease; Calcium Score; Radiotherapy; Cardiovascular events; CV risk factors; Cardio-oncology
MeSH Terms: conditions — Breast Neoplasms; Coronary Artery Disease | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Other): After signing the informed consent form, patients who meet all eligibility criteria will be enrolled in the Study. After execution of the CT scan the patient will be contacted to discuss the CT scan result. In case of high calcium score values, patients will be performing a cardiological medical examination, ECG, and further diagnostic investigations, as clinically indicated
  Interventions: Diagnostic Test: CT scan and blood sample collection

INTERVENTIONS:
Diagnostic Test: CT scan and blood sample collection — Each enrolled patient performs:
  * preventive clinical cardiology assessment visit, addressed to individualized risk profile assessment and addressed to chest CT scan.
  * a blood sampling (1 citrate tube of 5 ml) will be done the same day just the chest CT scan and analyzed locally also for future research of biomarker discovery (single sample, for those patients who agree in ICF)
  * CT scan

SUMMARY:
This is a no-profit, national, monocenter, retrospective, and prospective low-intervention study. It is a low-intervention study in terms of diagnostic additional procedure (CT scan). It is planned to recruit a maximum of 100 women diagnosed with early-stage breast cancer and treated with adjuvant breast radiotherapy from 2010 to 2017 at the European Institute of Oncology who meet all the inclusion and exclusion criteria. The aim of the Study is to analyze a population of breast cancer patients treated by adjuvant whole breast radiotherapy to identify the most important cardiovascular (CV) risk factors linked to coronary artery disease (CAD) development, in a cure-without-complications oncology strategy.

DETAILED DESCRIPTION:
In the present study a pre-screening activity is planned, that will be conducted by the European Institute of Oncology (IEO) at the Division of Radiotherapy. It will be done to identify and select from the IEO's database about 100 women diagnosed with early-stage breast cancer and treated with adjuvant breast radiotherapy, from 2010 to 2017, and with a > 5 years clinical Follow up (FU). All patients, who present pre-specified RT treatment, in terms of radiation exposure, and radiation protocol (IORT excluded as well as previous RT treatments), will be proposed to participate in the Study. The researcher of the IEO will contact by phone each identified patient (eligible patients) to request her interest in participating in the present study and to obtain her availability to be contacted by the Investigator of Centro Cardiologico Monzino (CCM) to define all aspects and activities planned in the protocol.

Patients who meet all eligibility criteria, after signing the informed consent form, at Centro Cardioogico Monzino, will be enrolled in the study. After execution of the CT scan the patient will be contacted to discuss the CT scan result. In case of high calcium score values, patients will be performing a cardiological medical examination, ECG, and further diagnostic investigations, as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with early-stage breast cancer treated with adjuvant whole breast external beam radiotherapy from 2010 to 2017;
* Patients with a > 5 years clinical follow-up (FU) from diagnosis of breast cancer
* Adult women/patients ≥18 years old and ≤ 60 years at time of radiation therapy;
* Patients with homogeneous and standardized radiation exposure protocol (external beam radiotherapy 40 Gy in 15 fractions)
* Patients who have signed the written informed consent

Exclusion Criteria:

* Patients aged < 18 or > 60 years at time of radiation therapy;
* Patients with bilateral breast cancer or breast cancer of unknown laterality;
* Patients with a prior diagnosis of invasive cancer (apart from non-melanoma skin cancer);
* Patients with known active ischemic heart disease during or before the RT period;
* Patients with no definitive surgery (e.g. a biopsy only);
* Patients who did not receive radiotherapy were excluded from the Study.
* Patients who are currently participating in an investigational interventional study.
* IORT (Intraoperative radiotherapy) and PBI (partial breast radiotherapy) excluded
* Participants not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to Study procedures

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women diagnosed with early-stage breast cancer and treated with adjuvant breast radiotherapy from 2010 to 2017 at European Institute of Oncology
Enrollment: 92 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Coronary calcium (CAC) | 2 years
  Coronary calcium (CAC) assessment and its relationship with left-side or right-side breast radiation therapy and previously known cardiovascular risk factors. The quantification of CAC will be performed according to the Agatston score by multiplying the total CAC area in mm2 by a density factor ranging from 1 to 4 (1 for lesions with a density of 130-199 HU; 2 if the lesion has a density of 200-299 HU; 3 for lesions with a density of 300-399 HU; 4 for densities ≥400 HU)

SECONDARY OUTCOMES:
Outcome 2 circulating markers | 2 years
  Evaluate circulating markers, mostly related to radiation-induced oxidative stress and correlate them to previous CV events and CT data obtained. Patients will undergo a blood sample withdrawal focused on evaluation of albumin isoforms in human plasma and protein signatures.
  Albumin thiolation: Mercaptoalbumin (HSA-SH) and thiolated albumin (+120 ± 2 Da, Thio-HSA) will be detected and their intensities used to calculate the relative abundances. Targeted Proteomics will be performed and relative quantitation will be expressed in Normalized protein expression (NPX), Normalized Protein eXpression, is Olink's arbitrary unit which is in Log2 scale. It is calculated from Ct values and data pre-processing (normalization) is performed to minimize both intra- and inter-assay variation. NPX data allows users to identify changes for individual protein levels across their sample set, and then use this data to establish protein signatures.
Outcome 3 Incidence of CV events | 2 years
  Incidence of CV events in relationship to left vs right-side breast radiation

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Trabattoni, MD, Principal Investigator — IRCCS Centro Cardiologico Monzino
Locations (1):
- IRCCS Centro Cardiologico Monzino, Milan, Italy

REFERENCES:
- [Derived] Trabattoni D, Leonardi MC, Mancini ME, Jereczek-Fossa BA, Cattani F, Santagostino Baldi G, Bonomi A, Galotta A, Mushtaq S, Annoni A, Alio D, Vincini MG, Fodor CI, La Grutta L, Montorsi P, Pontone G. Coronary artery calcium and cardiovascular risk factors analysis after radiotherapy for breast cancer (the CLARIFIER: a gender-based preventive medicine study). Front Cardiovasc Med. 2025 Aug 4;12:1615793. doi: 10.3389/fcvm.2025.1615793. eCollection 2025. PMID 40832141